CLINICAL TRIAL: NCT05932862
Title: An Open-Label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of XL309 (ISM3091) as Single-Agent and Combination Therapy in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of XL309 (ISM3091) Alone and in Combination in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL309-101
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
Keywords: Ovarian Cancer; Prostate Cancer; Pancreatic Cancer; Advanced HRRm Solid Tumors; Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation Single Agent Evaluation (Experimental): Participants will receive XL309 in sequential cohorts of increasing doses.
  Interventions: Drug: XL309
- Dose Escalation Combination Therapy (Experimental): Participants will receive XL309 in sequential cohorts of increasing doses in combination with olaparib.
  Interventions: Drug: XL309; Drug: Olaparib
- Cohort Expansion Stage Single Agent Evaluation (Experimental): The recommended dose as determined in the Escalation Stage will be further studied in advanced solid tumor-specific cohorts.
  Interventions: Drug: XL309
- Cohort Expansion Stage Combination Therapy Evaluation (Experimental): The recommended dose as determined in the Escalation Stage will be further studied in combination with olaparib in advanced solid tumor-specific cohorts.
  Interventions: Drug: XL309; Drug: Olaparib

INTERVENTIONS:
Drug: XL309 — XL309 will be administered orally per assigned schedule.
  Other Names: ISM3091
Drug: Olaparib — Olaparib will be administered orally per assigned schedule.
  Arms: Cohort Expansion Stage Combination Therapy Evaluation; Dose Escalation Combination Therapy

SUMMARY:
This is a first-in-human (FIH), multicenter, open-label Phase I study to investigate the safety, tolerability, preliminary antitumor activity, as well as pharmacokinetics (PK) and pharmacodynamics of XL309 (previously ISM3091) administered alone or in combination with olaparib in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Capable of understanding and complying with protocol requirements.
2. Male or female aged 18 years or older.
3. Eastern Cooperative Oncology Group performance status 0 or 1.
4. Adequate bone marrow and organ function.
5. Participant-disease Characteristics

   Dose-Escalation Stage Single Agent and Combination:

   a) Participants whose tumor progressed on, or who were intolerant to standard therapy, have a disease for which no therapy exists or are not a candidate for these therapies, and have one of the following cancers:

   i. Histologically confirmed locally advanced/metastatic human epidermal growth factor receptor-2 (HER2)-negative breast cancer, with deleterious or suspected deleterious breast cancer gene (BRCA)1/2 alteration.

   ii. Histologically confirmed locally advanced/metastatic high-grade serous ovarian cancer (HGSOC), including primary peritoneal cancer (PPC) and fallopian tube cancer (FTC).

   iii. Histologically confirmed locally advanced/metastatic CRPC, with deleterious or suspected deleterious BRCA1/2 alteration.

   iv. Histologically confirmed locally advanced/metastatic pancreatic cancer with deleterious or suspected deleterious BRCA1/2 alteration.

   v. Locally advanced/metastatic tumors with deleterious or suspected deleterious germline or somatic homologous recombination repair (HRR) mutation or homologous recombination deficiency (HRD) phenotype.

   Cohort-Expansion Stage Single Agent and Combination:

   b) HER2-negative breast cancer cohort: participants with histologically confirmed locally advanced/metastatic (HER2)-negative breast cancer with alterations in select HRR genes.

   c) Platinum-sensitive HGSOC cohort: participants with histologically confirmed locally advanced/metastatic HGSOC, including primary peritoneal cancer (PPC) and fallopian tube cancer (FTC), with positive HRD result using an approved diagnostic, and/or alterations in select HRR genes.

   d) mCRPC cohort: participants with metastatic, castration-resistant adenocarcinoma of the prostate with alterations in select HRR genes.

   e) HRRm advanced solid tumors cohort: participants with locally advanced/metastatic tumors with alterations in select HRR genes.

   For all participants with solid tumors:
6. Participants in the Cohort-Expansion Stage must have at least 1 measurable target lesion.
7. Recovery to baseline or ≤ Grade 1 CTCAE v5 from AE(s) related to any prior treatments.

Key Exclusion Criteria

1. Prior anticancer treatment including:

   1. Small molecule-targeted therapy < 5 half-lives from first dose of study treatment, or 3 weeks (whichever is shorter).
   2. Any antibody therapy < 5 half-lives from first dose of study treatment (or 4 weeks since last therapy, whichever is shorter).
   3. Chemotherapy with nitrosoureas or mitomycin C < 6 weeks from first dose of study treatment. Other chemotherapy < 3 weeks prior to first dose of study treatment.
   4. Radiation therapy (including radiofrequency ablation) < 1 week prior to initiation of study treatment. Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible.
2. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.
3. History of hypersensitivity to any excipient of XL309, or history of allergic reactions attributed to drugs with a similar chemical or biologic structure or class to XL309.
4. Lactating or pregnant females.
5. Clinically relevant cardiovascular disease.
6. Known history of myelodysplastic syndrome.
7. Other severe, acute, or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or that may interfere with the interpretation of the study results, and in the judgment of the investigator, would make the participant inappropriate for the study.
8. Inability or unwillingness to comply with requirement for oral drug administration or presence of a gastrointestinal condition that would preclude adequate absorption of XL309.
9. Prior treatment with a ubiquitin specific peptidase 1 (USP1) inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2029-01-03 (Estimated); Study Completion 2029-08-03 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Stage: Incidence of TEAEs and SAEs; AEs Leading to Dose Modification, Discontinuation, or Death; and Laboratory Abnormalities | Approximately 24 months
  Adverse events will be recorded and severity graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Dose Escalation Stage: Incidence of Dose-Limiting Toxicities (DLTs) | Approximately 24 months
Dose Escalation Stage: XL309 Exposure Over Time Measured as Area Under the Plasma Concentration Curve (AUC) | Approximately 24 months
Dose Escalation Stage: XL309 Maximum Plasma Concentration (Cmax) | Approximately 24 months
Dose Escalation Stage: XL309 Time to Cmax | Approximately 24 months
Dose Escalation Stage: XL309 Trough Concentration (Ctrough) | Approximately 24 months
  Lowest concentration of drug in the bloodstream, measured just before the next dose is administered.
Dose Escalation Stage: XL309 Apparent Clearance (CL/F) | Approximately 24 months
Cohort Expansion Stage: Incidence of TEAEs and SAEs; AEs Leading to Dose Modification, Discontinuation, or Death; and Laboratory Abnormalities | Approximately 24 months
  Adverse events will be recorded and severity graded using CTCAE version 5.0.
Cohort Expansion Stage: Objective Response Rate (ORR) | Approximately 24 months
  ORR will be measured per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as assessed by the Investigator. ORR for prostate cancer will be based on Prostate Cancer Working Group 3 (PCWG3) criteria, as assessed by the Investigator

SECONDARY OUTCOMES:
Dose Escalation Stage: Olaparib Exposure Over Time Measured as Area Under the Plasma Concentration Curve (AUC) at Steady State | Approximately 24 months
Dose Escalation Stage: Olaparib Cmax at Steady State | Approximately 24 months
Dose Escalation Stage: Olaparib Ctrough at Steady State | Approximately 24 months
Cohort Expansion Stage: Concentration of XL309 in Plasma at Specified Time Points | Approximately 24 months
Cohort Expansion Stage: Concentration of Olaparib in Plasma at Specified Time Points | Approximately 24 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Exelixis Clinical Site #12, Fountain Valley, California
  - Exelixis Clinical Site #15, Jacksonville, Florida
  - Exelixis Clinical Site #8, Orlando, Florida
  - Exelixis Clinical Site #16, Tampa, Florida
  - Exelixis Clinical Site #14, Rochester, Minnesota
  - Exelixis Clinical Site #10, Kansas City, Missouri
  - Exelixis Clinical Site #9, New Brunswick, New Jersey
  - Exelixis Clinical Site #5, New York, New York
  - Exelixis Clinical Site #7, Cleveland, Ohio
  - Exelixis Clinical Site #13, Oklahoma City, Oklahoma
  - Exelixis Clinical Site #11, Germantown, Tennessee
  - Exelixis Clinical Site #6, Nashville, Tennessee
  - Exelixis Clinical Site #4, Austin, Texas
  - Exelixis Clinical Site #1, Houston, Texas
  - Exelixis Clinical Site #2, Houston, Texas
  - Exelixis Clinical Site #3, San Antonio, Texas